CLINICAL TRIAL: NCT00005773
Title: Early Inhaled Nitric Oxide Therapy in Term and Near Term Infants With Respiratory Failure
Brief Title: Early Inhaled Nitric Oxide for Respiratory Failure in Newborns
Acronym: Early iNO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Halted after 3 years because of a persistent decline in enrollment
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); Mallinckrodt (Industry)
Responsible Party: G. Ganesh Konduri, Lead Principal Investigator, Medical College of Wisconsin, Children's Hospital of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0019; U01HD019897 (NIH); U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD021397 (NIH); U10HD021415 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027881 (NIH); U10HD027904 (NIH); U10HD034167 (NIH); U10HD034216 (NIH); U10HD040689 (NIH); M01RR000070 (NIH); M01RR000633 (NIH); M01RR000750 (NIH); M01RR000997 (NIH); M01RR001032 (NIH); M01RR006022 (NIH); M01RR008084 (NIH); M01RR016587 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Infant, Newborn; Hypertension, Pulmonary; Persistent Fetal Circulation Syndrome; Pneumonia, Aspiration; Respiratory Distress Syndrome, Newborn; Respiratory Insufficiency
Keywords: NICHD Neonatal Research Network; Hypertension, pulmonary; Hypoxic respiratory failure; Meconium aspiration; Methemoglobinemia; Nitric oxide; Oxygen inhalation therapy; Persistent Fetal Circulation Syndrome; Pneumonia, aspiration; Respiratory distress syndrome; Respiratory insufficiency; Severe respiratory failure
MeSH Terms: conditions — Hypertension, Pulmonary; Persistent Fetal Circulation Syndrome; Pneumonia, Aspiration; Respiratory Distress Syndrome, Newborn; Respiratory Insufficiency; Meconium Aspiration Syndrome; Methemoglobinemia; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early iNO Management (Experimental): Initiation of iNO in use for term and near-term infants in respiratory failure with an oxygenation index between 15-25.
  Interventions: Drug: Inhaled Nitric Oxide
- Standard iNO management (Active Comparator): Begin a sham initiation of iNO in term and near-term infants in respiratory failure with an oxygenation index (OI) between 15-25; initiated actual iNO therapy based on standard threshold (OI >=25).
  Interventions: Drug: Standard iNO therapy

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Study gas was initiated at a concentration of 5 ppm, and the dose was increased to 20 ppm when the infant had <=20 mm Hg increase in PaO2 (less than full response).
  Arms: Early iNO Management
Drug: Standard iNO therapy — Begin a sham initiation of iNO in term and near-term infants in respiratory failure with an oxygenation index (OI) between 15-25; initiated actual iNO therapy based on standard threshold (OI >=25).
  Arms: Standard iNO management

SUMMARY:
This prospective, randomized controlled trial tested whether initiating iNO therapy earlier would reduce death and reduce the use of extracorporeal membrane oxygenation (ECMO) -- temporary lung bypass -- therapy compared with the standard recommendation threshold. Infants who were born at >34 weeks' gestation were enrolled when they required assisted ventilation and had an oxygenation index (OI) >15 and <25 on any 2 measurements in a 12-hour interval. Infants were randomized to receive either early iNO or to simulated initiation of iNO (control). Infants who had an increase in OI to 25 or more were given iNO as standard therapy. The neurodevelopment of the subjects were evaluated at 18-22 months corrected age.

DETAILED DESCRIPTION:
Respiratory failure occurs in near term and term infants as a complication of perinatal aspiration syndromes, pneumonia, sepsis, respiratory distress syndrome and primary pulmonary hypertension. Recently a collaborative trial of the NICHD Neonatal Research Network and the Canadian Inhaled Nitric Oxide Study Group (the NINOS trial) demonstrated that inhaled nitric oxide (iNO) reduced the number of deaths and the need for extracorporeal membrane oxygenation (ECMO) therapy -- a lung bypass mechanism -- from 64 percent to 46 percent. The standard recommended threshold for initiation of iNO therapy, based on this trial, was an oxygenation index (OI) >=25.

The purpose of this study is to determine if administration of inhaled nitric oxide earlier in the course of respiratory failure and to infants with less severe respiratory failure, decreases the incidence of ECMO or death, as suggested by the sub-group analysis of the original NINOS trial. This prospective, randomized controlled trial tested whether initiating iNO therapy earlier would reduce death and reduce the use of ECMO therapy compared with the standard recommendation threshold.

Infants who were born at >34 weeks' gestation (near- or full-term) were enrolled when they required assisted ventilation and had an oxygenation index (OI) >15 and <25 on any 2 measurements in a 12-hour interval. Infants were randomized to receive either early iNO or to simulated initiation of iNO (control). Infants who had an increase in OI to 25 or more were given iNO as standard therapy. The neurodevelopment of the subjects were evaluated at 18-22 months corrected age.

The study compared the outcome of infants received iNO at OI >15 and <25, with a control group that received a simulated early procedure with iNO actually given based on the standard recommendation. iNO was delivered at 20 ppm during the initial dose-response evaluation. Infants in either group who showed subsequent deterioration with OI >25 on two consecutive measurements at least one hour apart, or a rapid deterioration with OI >30 on two consecutive measurements 15 minutes apart, received iNO therapy as part of standard medical management. Specific guidelines were followed for the use of high frequency ventilation and surfactant during study gas administration to prevent them from confounding the results of the study.

Study recruitment was discontinued after 3 years due to a persistent decline in enrollment.

Infants were given neurodevelopmental exams at 18-22 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at >34 weeks gestational age
* Require assisted ventilation for hypoxic respiratory failure
* Have a diagnosis of primary persistent pulmonary hypertension (PPHN), respiratory distress syndrome, perinatal aspiration syndrome, pneumonia/sepsis, or suspected pulmonary hypoplasia
* Have an oxygenation index >15 and <25 based on 2 arterial blood gases taken at least 15 minutes apart or an Fi02 >80%
* In-dwelling arterial line
* Parental consent

Exclusion Criteria:

* Known structural congenital heart disease, except patent ductus arteriosus and atrial level shunts
* Congenital diaphragmatic hernia
* Use of high frequency jet ventilation at the time of randomization
* Prior exposure to inhaled nitric oxide therapy

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 1998-08; Primary Completion 2001-05 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Death or use of extracorporeal membrane oxygenation (ECMO) | Hospital discharge or 120 days of life

SECONDARY OUTCOMES:
Use of iNO therapy based on the standard recommended threshold | Hospital Discharge or 120 days of life
Progression to severe respiratory failure (OI>40) | Hospital discharge or 120 days of life
  Severe respiratory failure, defined as OI >40
Neurodevelopmental impairment | 18-22 months corrected age

CONTACTS AND LOCATIONS:
Overall Officials: G. Ganesh Konduri, MD, Study Director — University of Wisconsin, Madison; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Carlos Fajardo, MD, Principal Investigator — St. Joseph's Hospital; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Gail Knight, MD, Principal Investigator — San Diego Children's Hospital; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Charles R. Bauer, MD, Principal Investigator — University of Miami; Barbara J. Stoll, MD, Principal Investigator — Emory University; Greg M. Sokol, MD, Principal Investigator — Indiana University; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Avroy A. Fanaroff, MD, Study Director — Case Western Reserve University, Rainbow Babies and Children's Hospital; William Oh, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Abbot R. Laptook, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Mary Wearden, MD, Principal Investigator — Baylor College of Medicine; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Dennis E. Mayock, MD, Principal Investigator — University of Washington
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - San Diego Children's Hospital, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Washington School of Medicine, Seattle, Washington

REFERENCES:
- [Background] Sokol GM, Van Meurs KP, Wright LL, Rivera O, Thorn WJ 3rd, Chu PM, Sams RL. Nitrogen dioxide formation during inhaled nitric oxide therapy. Clin Chem. 1999 Mar;45(3):382-7. PMID 10053039
- [Background] Sokol GM, Ehrenkranz RA. Inhaled nitric oxide therapy in neonatal hypoxic respiratory failure: insights beyond primary outcomes. Semin Perinatol. 2003 Aug;27(4):311-9. doi: 10.1016/s0146-0005(03)00043-0. PMID 14510322
- [Result] Konduri GG, Solimano A, Sokol GM, Singer J, Ehrenkranz RA, Singhal N, Wright LL, Van Meurs K, Stork E, Kirpalani H, Peliowski A; Neonatal Inhaled Nitric Oxide Study Group. A randomized trial of early versus standard inhaled nitric oxide therapy in term and near-term newborn infants with hypoxic respiratory failure. Pediatrics. 2004 Mar;113(3 Pt 1):559-64. doi: 10.1542/peds.113.3.559. PMID 14993550
- [Result] Konduri GG, Vohr B, Robertson C, Sokol GM, Solimano A, Singer J, Ehrenkranz RA, Singhal N, Wright LL, Van Meurs K, Stork E, Kirpalani H, Peliowski A, Johnson Y; Neonatal Inhaled Nitric Oxide Study Group. Early inhaled nitric oxide therapy for term and near-term newborn infants with hypoxic respiratory failure: neurodevelopmental follow-up. J Pediatr. 2007 Mar;150(3):235-40, 240.e1. doi: 10.1016/j.jpeds.2006.11.065. PMID 17307536
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/